CLINICAL TRIAL: NCT04334798
Title: Effectiveness of Different Modalities of Motor Learning of Pelvic Floor Muscle Contraction in Women With Pelvic Floor Dysfunction: Randomized Controlled Trial
Brief Title: Pelvic Floor Consciousness in Women With Pelvic Floor Dysfunction
Acronym: PFMCON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Maria Torres Lacomba, Principal investigator & Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OE14/2020
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Pelvic Floor Disorders
Keywords: Motor Learning; Pelvic Floor Muscles; Physiotherapy; Biofeedback; Consciousness
MeSH Terms: conditions — Pelvic Floor Disorders | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PFM&electro&BFB (Experimental): An educational program (anatomical and physiological explanation of the abdomen-pelvic cavity (perineal organs, bone, ligament and muscle structures of the entire abdomen-pelvic cavity; knack) will be implemented, and active exercises of the pelvic floor muscles (PFM) will be performed using intravaginal palpation and electrostimulation, together with biofeedback (BFB).
  Interventions: Other: Active exercises of the pelvic floor muscles & Electrostimulation & Biofeedback
- PFM&BFB (Experimental): An educational program (anatomical and physiological explanation of the abdomen-pelvic cavity (perineal organs, bone, ligament and muscle structures of the entire abdomen-pelvic cavity; knack) will be implemented, and active exercises of the PFM will be performed using intravaginal palpation together with biofeedback (BFB).
  Interventions: Other: Active exercises of the pelvic floor muscles & Biofeedback
- PFM&electro&transabdominal US (Experimental): An educational program (anatomical and physiological explanation of the abdomen-pelvic cavity (perineal organs, bone, ligament and muscle structures of the entire abdomen-pelvic cavity; knack) will be implemented, and active exercises of the PFM will be performed using intravaginal palpation and electrostimulation, together with transabdominal ultrasound biofeedback (BFB).
  Interventions: Other: Active exercises of the pelvic floor muscles & Electrostimulation &Transabdominal US Biofeedback
- PFM&transabdominal US (Experimental): An educational program (anatomical and physiological explanation of the abdomen-pelvic cavity (perineal organs, bone, ligament and muscle structures of the entire abdomen-pelvic cavity; knack) will be implemented, and active exercises of the PFM will be performed using intravaginal palpation together with transabdominal ultrasound biofeedback (BFB).
  Interventions: Other: Active exercises of the pelvic floor muscles & Transabdominal US Biofeedback

INTERVENTIONS:
Other: Active exercises of the pelvic floor muscles & Electrostimulation & Biofeedback — See information included in arm/group descriptions.
  Arms: PFM&electro&BFB
Other: Active exercises of the pelvic floor muscles & Biofeedback — See information included in arm/group descriptions.
  Arms: PFM&BFB
Other: Active exercises of the pelvic floor muscles & Transabdominal US Biofeedback — See information included in arm/group descriptions.
  Arms: PFM&transabdominal US
Other: Active exercises of the pelvic floor muscles & Electrostimulation &Transabdominal US Biofeedback — See information included in arm/group descriptions.
  Arms: PFM&electro&transabdominal US

SUMMARY:
The purpose of the study is to compare the efficacy of different modalities of motor learning of pelvic floor muscle contraction in women with pelvic floor dysfunctions, considering the efficacy of the treatment as improving the specific quality of life related to pelvic floor dysfunctions and improvement of the muscular properties of the pelvic floor muscles.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with pelvic floor dysfunction by their doctor.
* Women who are unable to voluntarily contract the pelvic floor muscles, quantified by the Modified Oxford Score by a score less than or equal to 2.

Exclusion Criteria:

* Women who are pregnant or women who have had a vaginal or caesarean birth in the past six months.
* Women whose PFD is severe, and the first indication is surgical (POP-Q grade III-IV prolapses).
* Women with pain in the pelvic-perineal region of 3 cm in the visual analog scale, where a score of 0 cm means no pain, and a score of 10 cm, the maximum pain that the participant can imagine.
* Women who have received pelvic floor physiotherapy treatment in the last 12 months.
* Women with any pathology that may affect the treatment (neurological, gynecological or urological), or with recurrent urinary infection or hematuria.
* Women with cognitive limitations to understand the information, answer the questionnaires, consent and / or participate in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in life impact of pelvic floor dysfunction | 5 assessments to evaluate change from baseline: at baseline, after the intervention period (2 months from baseline), 3 months, 6 months and 12 months after the intervention.
  It will be assessed by the Pelvic Floor Impact Questionnaire-7 (PFIQ-7) Spanish version. The PFIQ-7 consists of 3 scales of 7 questions each taken from the Urinary Impact Questionnaire, the Pelvic Organ Prolapse Impact Questionnaire, and the Colorectal-Anal Impact Questionnaire. The 3 scales are scored from 0 (least impact) to 100 (greatest impact) and an overall summary score (0 to 300).
Change in symptoms and quality of life | 5 assessments to evaluate change from baseline: at baseline, after the intervention period (2 months from baseline), 3 months, 6 months and 12 months after the intervention.
  It will be assessed by the Pelvic Floor Distress Inventory-20 (PFDI-20) Spanish version that is both a symptom inventory and a measure of the degree of bother and distress caused by pelvic floor symptoms. The PFDI-20 includes 20 questions and 3 scales. Each of the 3 scales is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 - 300 and the higher the score, the worse quality of life. The 3 scales include questions taken from the following widely used outcome measures: Urinary Distress Inventory - 6 questions, Pelvic Organ Prolapse (POP) Distress Inventory - 6 questions, and Colorectal-Anal Distress Inventory - 8 questions collecting data about Urinary Incontinence (UI), POP and colorectal and anal symptoms.

SECONDARY OUTCOMES:
Change in pelvic floor muscle strength by manual scale | 5 assessments to evaluate change from baseline, after the intervention period (2 months from baseline), 3 months, 6 months and 12 months after the intervention.
  It will be measured by Modified Oxford Scale to rate pelvic floor muscle contraction on a scale of 0-5: 0 = no contraction; 1 = minor muscle; 'flicker'; 2 = weak muscle; contraction; 3 = moderate muscle contraction; 4 = good muscle contraction and 5 = strong muscle contraction.
Change in pelvic floor muscle strength by dynamometry | 5 assessments to evaluate change from baseline, after the intervention period (2 months from baseline), 3 months, 6 months and 12 months after the intervention.
  It will be measured by dynamometry (measured in GRAMS).
Change in pelvic floor muscle passive tone | 5 assessments to evaluate change from baseline, after the intervention period (2 months from baseline), 3 months, 6 months and 12 months after the intervention.
  It will be measured by dynamometry (measured in GRAMS).
Change in the displacement of the base of the bladder during voluntary contraction of the pelvic floor | 5 assessments to evaluate change from baseline, after the intervention period (2 months from baseline), 3 months, 6 months and 12 months after the intervention.
  It will be measured by Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: María Torres-Lacomba, PhD, Principal Investigator — University of Alcalá
Locations (3):
- Spain (3):
  - Physiotherapy in women´s health research group. University of Alcalà, Alcalà de Henares, Madrid
  - María Torres-Lacomba, Alcalá de Henares, Madrid
  - University of Alcalá. FPSM research group. HUPA, Alcalá de Henares, Madrid

IPD SHARING:
Plan to Share IPD: No